CLINICAL TRIAL: NCT00471328
Title: A Randomized, Open-label, Multi-center Study to Evaluate the Efficacy of Nilotinib Versus Best Supportive Care With or Without a Tyrosine Kinase Inhibitor (Investigator's Choice) in Adult Patients With Gastrointestinal Stromal Tumors Resistant to Both Imatinib and Sunitinib
Brief Title: Efficacy and Safety of Nilotinib (AMN107) Compared With Current Treatment Options in Patients With GIST Who Have Failed Both Imatinib and Sunitinib
Acronym: ENEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2201; 2006-002267-11 (EudraCT Number); NCT00488150 (obsolete NCT alias)
Record Dates: First submitted 2007-04-26; First posted 2007-05-09 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; adults; imatinib resistant; sunitinib resistant; AMN107; nilotinib; treatment; Gastrointestinal stromal tumor (GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib; Imatinib Mesylate; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib (Experimental): 400mg twice daily in core and extension phases of the study.
  Interventions: Drug: Nilotinib
- Control/cross-over to Nilotinib (Active Comparator): In core study phase, patients in this arm received Best Supportive Care (BSC) with or without imatinib or sunitinib at the last tolerated dose or at the investigator's choice until documented disease progression followed by cross-over to nilotinib arm.
  Patients entering the extension study on this control arm were permitted to cross over to nilotinib arm only upon documented disease progression.
  Interventions: Drug: Nilotinib; Other: Best Supportive Care (BSC) +/- imatinib or sunitinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 400 mg twice daily (bid)
  Other Names: AMN107, Tasigna®
Other: Best Supportive Care (BSC) +/- imatinib or sunitinib — Can include pain medication, localized radiotherapy, nutritional support, and/or oxygen therapy and blood transfusions. Imatinib or sunitinib can be administered at the last tolerated dose and regimen or at the Investigator's choice.
  Arms: Control/cross-over to Nilotinib

SUMMARY:
The study evaluated the safety and efficacy of nilotinib versus current treatment in adults with gastrointestinal stromal tumors (GIST) who have either progressed or who were intolerant to the first and second line treatments.

ELIGIBILITY:
Inclusion criteria (Core Phase):

* Age ≥18 years
* Radiological confirmation of disease progression during imatinib and sunitinib therapy OR intolerance to imatinib and/or sunitinib
* At least one measurable site of disease on CT/MRI scan
* Physically fit even if not able to work
* Normal organ, electrolyte, and bone marrow function

Inclusion criteria (Extension Phase):

* Patients whose tumors had progressed on the control arm and had crossed over to the nilotinib arm.
* The study was stopped due to meeting the primary efficacy endpoint of PFS at the interim analysis.
* Patients who were still being treated at the close of the Core study on the control arm or nilotinib arm (whose tumors have not progressed at the time of the end of the Core study).
* Patients must have had documented, confirmed stable, partial or complete response as defined by the RECIST criteria at the time of entry into the Extension study with the exception of patients who had progressed on the control arm.

Exclusion criteria (Core Phase):

* Previous treatment with nilotinib or any other drug in this class or other targeted therapy
* Treatment with any cytotoxic and/or investigational cytotoxic drug ≤ 4 weeks prior to study entry
* Impaired cardiac function
* Use of coumarin derivatives (i.e. warfarin, acenocoumarol, phenprocoumon)
* Women who are pregnant or lactating

Exclusion criteria (Extension Phase):

* Use of other anticancer treatments or investigational drugs (with exception of the study drugs)
* Patients with a history of noncompliance with study drug treatment in the Core study protocol.

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (11):
  - UCLA's Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Washington Hospital Center - Washington Cancer Institute, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Hospital, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Wertz Clinical Cancer Center, Detroit, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, East Melbourne, Victoria
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Toronto, Canada
- Novartis Investigative Site, Prague, Czechia
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
- Italy (2):
  - Novrtis Investigative Site, Bologna
  - Novartis Investigative Site, Milan
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Madrid, Spain
- Novartis Investigative Site, Chur, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients ongoing on treatment at primary analysis had option to enter extension. Patients in control arm were allowed cross over to Nilotinib arm at disease progression and considered as part of extension. Patients entering the extension part on control arm were permitted to cross over to the nilotinib only upon documented disease progression.
Groups:
- Nilotinib: 400 mg was taken orally twice daily in core and extension phase of the study
- Control/Cross Over to Nilotinib: In core study phase, patients in this arm received Best Supportive Care (BSC) with or without imatinib or sunitinib at the last tolerated dose or at the investigator's choice until documented disease progression followed by cross-over to nilotinib arm.
  Patients entering the extension study on this control arm were permitted to cross over to nilotinib arm only upon documented disease progression.
Period: Core Phase
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib
Started | 165 | 83
Crossover to Nilotinib:Started Extension | 0 | 53
Completed | 58 (Ongoing on treatment during completion of core.) | 16 (Ongoing on treatment during completion of core)
Not Completed | 107 | 67
Not completed — Adverse Event | 18 | 6
Not completed — Death | 8 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Abnormal laboratory value | 1 | 0
Not completed — Disease Progression | 78 | 53
Not completed — Administrative Problem | 0 | 1
Not completed — Protocol Deviation | 0 | 1
Period: Extension Phase
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib
Started | 41 (Out of 58 ongoing patients, 17 patients had progression or died before they could enter extension) | 67
Started:CrossOver Before PrimaryAnalysis | 0 | 53
Started:CrossOver After PrimaryAnalysis | 0 | 4
Started:CrossOver During Extension | 0 | 10
Completed | 0 | 0
Not Completed | 41 | 67
Not completed — Adverse Event | 3 | 12
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 1 | 7
Not completed — Protocol Deviation | 3 | 1
Not completed — Treatment duration as per protocol | 0 | 1
Not completed — Disease Progression | 32 | 44
Not completed — New cancer Therapy | 1 | 0
Not completed — Administrative Problem | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib | Total
Number analyzed (Participants) | 165 | 83 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 118 | 57 | 175
  >=65 years | 47 | 26 | 73
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.69) | 58.6 (10.57) | 57.8 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 36 | 100
  Male | 101 | 47 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 11 | 32
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 2 | 4 | 6
  White | 134 | 67 | 201
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) From Central Radiology Review Based on Primary Analysis (Data Cut-off: June, 2008)
Description: Progression-free survival (PFS) is the time from date of randomization to the date of first documented progression or death due to any cause. If a participant has not had an event, progression-free survival is censored at the time of last adequate tumor assessment. Progression is defined according to Modified Response Evaluation Criteria in Solid Tumors (modified RECIST) criteria as at least a 20% increase in the sum of the longest diameter of target lesions, worsening of the non-target lesions or the appearance of one or more new lesions.
Time Frame: Up to 16 months
Population: The intent to treat (ITT) population was defined as all randomized patients and was used as the primary efficacy population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 165 | 83
days | 109.0 [61.0 to 113.0] | 111.0 [60.0 to 116.0]

2. Secondary Outcome: Overall Survival Based on Primary Analysis (Data Cut-off:June, 2008)
Description: Overall survival (OS) is defined as the time from date of randomization to date of death due to any cause. If a participant is not known to have died, survival will be censored at the date of last contact.
Time Frame: Up to 16 months
Population: The intent to treat (ITT) population was defined as all randomized participants and was used as the primary efficacy population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 165 | 83
days | 332.0 [246.0 to NA] — The upper limit of CI was not computable due to insufficient number of events. | 280.0 [240.0 to 372.0]

3. Secondary Outcome: Overall Survival During Core and Extension Phases of the Study
Description: Overall survival (OS) is defined as the time from date of randomization to date of death due to any cause. If a participant is not known to have died, survival will be censored at the date of last contact. This analysis included both Core and Extension data as well as survival follow up data.
Time Frame: Up to 50 months (including core, extension and follow up period)
Population: Core Full Analysis Set (Core FAS): included all randomized patients included in the Core study. Analyses based on Core FAS does not account for treatment crossover i.e.pooling all data both before and after crossover. This analysis set was used to conduct an overall survival analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 165 | 83
days | 361 [265 to 425] | 300 [246 to 386]

4. Secondary Outcome: Overall Survival for Treatment Crossover Analysis Set
Description: For patients who crossed-over to nilotinib from the control arm, the overall survival was the time from the first dose date of nilotinib after switching from control arm to the date of death due to any cause. If death was not observed, the OS was censored at the latest date the patient was known to be alive.
Time Frame: Up to 34 months
Population: Treatment Crossover Analysis Set: All patients who crossed over from control arm to nilotinib after completing the Core study or during the Extension study after disease progression.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Control/Cross Over to Nilotinib: In core study phase, patients in this arm received Best Supportive Care (BSC) with or without imatinib or sunitinib at the last tolerated dose or at the investigator's choice until documented disease progression and cross-overed to nilotinib arm.
  Patients entering the extension study on this control arm were permitted to cross over to nilotinib arm only upon documented disease progression.
Arm/Group | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 67
days | 231 [196 to 327]

5. Primary Outcome: Progression-free Survival (PFS) From Local Investigator's Assessment Based on Treatment Crossover Analysis Set
Description: PFS is defined as the time from the first date of cross-over to nilotinib therapy from the control arm to the date of the first observation of documented disease progression. Tumor assessment was based on the local investigator's measurement using Modified Response Evaluation Criteria in Solid Tumors (modified RECIST) criteria. Progression is defined according to modified RECIST criteria as at least a 20% increase in the sum of the longest diameter of target lesions, worsening of the non-target lesions or the appearance of one or more new lesions.
Time Frame: Up to 34 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 67
days | 84 [56 to 109]

6. Secondary Outcome: Number of Responders With Confirmed Best Overall Response of Complete Response (CR) or Partial Response (PR) From Central Radiology Review During Primary Analysis (Data Cut-off: June, 2008)
Description: The best overall response is the best response recorded from randomization until disease progression. The CR/PR must be confirmed by at least two determinations at least 4 weeks apart before progression. Using modified RECIST criteria, a Complete Response is defined as disappearance of all lesions, and a Partial Response is defined as either 1) at least a 30% decrease in the sum of the longest diameter of target lesions and no new lesions or progression of non-target lesions or 2) disappearance of all target lesions but persistence of one or more non-target lesion(s).
Time Frame: Up to 16 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 165 | 83
Participants | 1 [0.0 to 3.3] | 0 [0.0 to 0.0]

7. Secondary Outcome: Number of Responders With Confirmed Best Overall Response of Complete Response (CR) or Partial Response (PR) From Local Investigator's Assessment Based on Treatment Crossover Analysis Set
Description: The best overall response (CR/PR) must be confirmed by at least two determinations at least 4 weeks apart before progression. Using modified RECIST criteria, a Complete Response is defined as disappearance of all lesions, and a Partial Response is defined as either 1) at least a 30% decrease in the sum of the longest diameter of target lesions and no new lesions or progression of non-target lesions or 2) disappearance of all target lesions but persistence of one or more non-target lesion(s).
Time Frame: Up to 34 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 67
Participants | 1 [0.0 to 8.0]

8. Secondary Outcome: Overall Clinical Benefit (Complete Response [CR]/Partial Response [PR] or Stable Disease [SD]) From Central Radiology Review Based on Primary Analysis (Data Cut-off: June, 2008)
Description: The overall clinical benefit includes the best overall responses of CR, PR, or SD. The best overall responses of CR/PR must be confirmed by at least two determinations at least 4 weeks apart before progression. The best overall response of SD must have at least one SD (or better) at least 6 weeks (or 6 months or 12 months as applicable) after randomization but before progression.
Time Frame: Up to 16 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nilotinib | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 165 | 83
Percentage of Participants
  CR/PR/SD | 52.7 [44.8 to 60.5] | 44.6 [33.7 to 55.9]
  CR/PR/SD lasting > 6 months | 7.3 [3.8 to 12.4] | 1.2 [0.0 to 6.5]
  CR/PR/SD lasting > 12 months | 0.6 [0.0 to 3.3] | 0 [0 to 0]

9. Secondary Outcome: Overall Clinical Benefit (Complete Response [CR]/Partial Response [PR] or Stable Disease [SD]) From Local Investigator's Assessment Based on Treatment Crossover Analysis Set
Description: as for outcome 8
Time Frame: Up to 34 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control/Cross Over to Nilotinib
Number analyzed (Participants) | 67
Percentage of Participants
  CR/PR/SD | 37.3 [25.8 to 50.0]
  CR/PR/SD lasting > 6 months | 7.5 [2.5 to 16.6]
  CR/PR/SD lasting > 12 months | 6.0 [1.7 to 14.6]

ADVERSE EVENTS:
Groups:
- Nilotinib(Core +Extension): Patients randomized to 400 mg Nilotinib which was taken orally twice daily. The safety is assessed using these patient's data from both core and extension phase of the study.
- Control(Core + Extension): Patients randomized to control arm, Best Supportive Care (BSC) with or without imatinib or sunitinib at the last tolerated dose before the study or at the dose of the investigator's choice. The safety is assessed using these patient's data from both core and extension phase of the study.
- Crossover Nilotinib Therapy: All patients who crossed over from control arm to nilotinib after completing the Core study or during the Extension study after disease progression were included in safety assessment.
Arm/Group | Nilotinib(Core +Extension) | Control(Core + Extension) | Crossover Nilotinib Therapy
Serious Adverse Events (participants affected / at risk) | 81/165 | 27/83 | 32/67
Other Adverse Events (participants affected / at risk) | 159/165 | 73/83 | 58/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib(Core +Extension) (N=165) | Control(Core + Extension) (N=83) | Crossover Nilotinib Therapy (N=67)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0
Spinocerebellar ataxia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 21 | 5 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 2 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 3 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 9 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 16 | 3 | 10
Generalised oedema (General disorders) | 0 | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 3
Pain (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 5 | 2 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Perihepatic abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 2
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Inferior vena caval occlusion (Vascular disorders) | 0 | 0 | 1
Intra-abdominal haemorrhage (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib(Core +Extension) (N=165) | Control(Core + Extension) (N=83) | Crossover Nilotinib Therapy (N=67)
Anaemia (Blood and lymphatic system disorders) | 39 | 17 | 12
Neutropenia (Blood and lymphatic system disorders) | 1 | 7 | 0
Eyelid oedema (Eye disorders) | 3 | 7 | 0
Abdominal distension (Gastrointestinal disorders) | 17 | 6 | 5
Abdominal pain (Gastrointestinal disorders) | 61 | 19 | 13
Abdominal pain lower (Gastrointestinal disorders) | 3 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 21 | 6 | 8
Ascites (Gastrointestinal disorders) | 3 | 5 | 3
Constipation (Gastrointestinal disorders) | 41 | 9 | 10
Diarrhoea (Gastrointestinal disorders) | 28 | 20 | 5
Dyspepsia (Gastrointestinal disorders) | 13 | 6 | 1
Nausea (Gastrointestinal disorders) | 51 | 33 | 13
Stomatitis (Gastrointestinal disorders) | 13 | 4 | 1
Vomiting (Gastrointestinal disorders) | 33 | 25 | 14
Asthenia (General disorders) | 46 | 6 | 9
Fatigue (General disorders) | 46 | 15 | 12
Oedema peripheral (General disorders) | 30 | 26 | 13
Pyrexia (General disorders) | 31 | 7 | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 14 | 1 | 4
Alanine aminotransferase increased (Investigations) | 14 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 12 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 15 | 4 | 1
Lipase increased (Investigations) | 11 | 0 | 1
Weight decreased (Investigations) | 34 | 7 | 20
Decreased appetite (Metabolism and nutrition disorders) | 47 | 18 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 5 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 4 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5
Dysgeusia (Nervous system disorders) | 9 | 1 | 0
Headache (Nervous system disorders) | 34 | 8 | 4
Insomnia (Psychiatric disorders) | 13 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 11 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Erythema (Skin and subcutaneous tissue disorders) | 10 | 1 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 26 | 7 | 4
Hypertension (Vascular disorders) | 8 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.